CLINICAL TRIAL: NCT07337772
Title: Prospective Randomized Controlled Trial Comparing Different Doses of Corticosteroids in Local Infiltration Analgesia (LIA) for Total Knee Arthroplasty
Brief Title: Comparing Different Doses of Corticosteroids in Local Infiltration Analgesia (LIA) for Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QT2025013-ZX
Record Dates: First submitted 2025-12-15; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Adrenal Cortex Hormones; Arthroplasty, Replacement, Knee; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-dose group (Experimental): LIA with the addition of 3 vials of Diprospan (each vial contains betamethasone 5 mg + betamethasone dipropionate 2 mg)
  Interventions: Drug: LIA with different doses of Diprospan
- Medium-dose group (Experimental): LIA with the addition of 2 vials of Diprospan (each vial contains betamethasone 5 mg + betamethasone dipropionate 2 mg)
  Interventions: Drug: LIA with different doses of Diprospan
- Low-dose group (Experimental): LIA with the addition of 1 vial of Diprospan (each vial contains betamethasone 5 mg + betamethasone dipropionate 2 mg)
  Interventions: Drug: LIA with different doses of Diprospan
- Control group (No Intervention): LIA without the addition of Diprospan

INTERVENTIONS:
Drug: LIA with different doses of Diprospan — LIA with different doses of Diprospan
  Arms: High-dose group; Low-dose group; Medium-dose group

SUMMARY:
This study aims to compare the efficacy of different doses of glucocorticoids in local infiltration analgesia (LIA) during total knee arthroplasty (TKA) through a prospective single-center randomized controlled trial, and to explore the safety and feasibility of high-dose glucocorticoids. Through this research, the investigators hope to provide an optimized solution for post-TKA pain management, improve patients' postoperative recovery and quality of life, and offer scientific evidence for pain management following TKA.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older;
2. Undergoing primary unilateral total knee arthroplasty (TKA)for unilateral knee osteoarthritis(OA)at ourhospital;
3. Preoperative American Society of Anesthesiologists(ASA)physical status classification of 1-3;
4. Ability to provide informed consent and sign a written informed consent form.

Exclusion Criteria:

1. Previous surgery on the operative knee or a history of infection in the operative knee;
2. Non-osteoarthritis conditions (including rheumatoid arthritis, traumatic arthritis, septic arthritis, and hemophilic arthritis);
3. Severe osteoarthritis (including flexion contracture >30° or varus/valgus deformity >30°);
4. Allergy to the relevant study drugs;
5. Presence of neuromuscular dysfunction in the ipsilateral limb;
6. Dependence on anesthetic drugs (defined as weekly use of opioids exceeding 100 mg morphine equivalents or local anesthetics for preoperative pain control for more than 3 months);
7. Poor systemic condition, including but not limited to: glycated hemoglobin (HbA1c) level >12%; blood pressure >170/110 mmHg (1 mmHg = 0.133 kPa); history of myocardial infarction, stroke, transient ischemic attack, acute congestive heart failure, or any acute coronary event within 6 months; dialysis or renal transplantation; pregnancy or lactation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Pain Score | Preoperatively (baseline), and at 6 hours, 12 hours, 24 hours, 48 hours, 3 weeks, and 6 weeks postoperatively.
  VAS ranges from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score | Preoperatively, and at 3 weeks and 6 weeks postoperatively.
  Patient-reported outcome measuring pain, stiffness, and physical function in knee osteoarthritis. Total score ranges from 0 (best) to 96 (worst). Lower scores indicate better outcomes.
range of motion | Preoperatively, and at 3 weeks and 6 weeks postoperatively.
  The range of motion (flexion and extension) of the operated knee will be measured using a standard goniometer. The primary outcome is the maximum active flexion angle (in degrees). A greater range of motion indicates better functional recovery.
Total Postoperative Analgesic Consumption | Within the first 48 hours postoperatively
  The total consumption of all analgesic medications administered for postoperative pain control. All doses will be converted to morphine milligram equivalents (MME) for opioids (e.g.,tramadol) and to standardized dosages for non-opioid analgesics (e.g., ibuprofen, celecoxib, acetaminophen). The outcome will be reported as total MME (for opioids) and total standardized dosage (for non-opioids), both as continuous measures.
. C-reactive Protein (CRP) Concentration | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Serum CRP level measured in milligrams per liter (mg/L). A key marker of systemic inflammation.
Erythrocyte Sedimentation Rate (ESR) | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Erythrocyte sedimentation rate measured in millimeters per hour (mm/h). A nonspecific marker of inflammation.
interleukin-6(IL-6) | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Serum IL-6 level measured in picograms per milliliter (pg/mL). A pro-inflammatory cytokine.
Alanine Aminotransferase (ALT) Concentration | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Serum ALT level measured in units per liter (U/L). Elevated levels may indicate liver injury.
Aspartate Aminotransferase (AST) Concentration | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Serum AST level measured in units per liter (U/L). Elevated levels may indicate liver or muscle injury.
Serum Creatinine Concentration | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Serum creatinine level measured in micromoles per liter (μmol/L). Elevated levels may indicate impaired renal function.
Blood Urea Nitrogen (BUN) Concentration | Postoperative Day 1, Day 4, Week 3, and Week 6.
  Blood urea nitrogen level measured in millimoles per liter (mmol/L). Elevated levels may be associated with dehydration or renal dysfunction.
Incidence of Local Complications | 0-6 months postoperatively
  The incidence of postoperative local complications at the surgical site, including but not limited to: wound exudation, poor wound healing, and periprosthetic joint infection. Incidence is defined as the number of participants experiencing at least one local complication, divided by the total number of participants in each group, expressed as a percentage.
Incidence of Systemic Complications | 0-6 months postoperatively
  The incidence of postoperative systemic complications, including but not limited to: nausea, vomiting, deep vein thrombosis (DVT), and acute liver failure. Incidence is defined as the number of participants experiencing at least one systemic complication, divided by the total number of participants in each group, expressed as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No